CLINICAL TRIAL: NCT03100604
Title: Prospective, Single-blind Study Investigating the Effect of Sevoflurane and Desflurane, Agents Used in Patients on the MEP
Brief Title: The Effect of General Anesthesia on the Middle Ear Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Sevtap Hekimoglu Sahin, Clinical Professor, Trakya University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013/136
Record Dates: First submitted 2016-08-31; First posted 2017-04-04 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Ear Deformities, Acquired
Keywords: middle ear pressure; sevoflurane; desflurane
MeSH Terms: conditions — Ear Deformities, Acquired | interventions — Desflurane; Sevoflurane

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- sevoflurane 2%, 1 MAC (Experimental): Maintenance of anesthesia was provided with 2% sevoflurane in S Group, and 6-9% desflurane in D Group, with 50% air /oxygen mixture and fresh gas flow at 4 l/min in both groups.
  Interventions: Drug: Sevoflurane
- Desfluran 6-9% 1MAC (Experimental): Maintenance of anesthesia was provided with 2% sevoflurane in S Group, and 6-9% desflurane in D Group, with 50% air /oxygen mixture and fresh gas flow at 4 l/min in both groups.
  Interventions: Drug: desflurane,

INTERVENTIONS:
Drug: desflurane, — Patients were divided into two groups according to inhalation agent administered for the surgery; Sevofluran, Group S (n=25) and Desfluran, Group D (N=25).
  Other Names: suprane
  Arms: Desfluran 6-9% 1MAC
Drug: Sevoflurane — For a drug, use generic name if established. Use the same name as in the associated Arm/Group Description(s).
  Other Names: sefoflurane
  Arms: sevoflurane 2%, 1 MAC

SUMMARY:
The investigators aimed to examine the effect of sevoflurane and desflurane, agents used in patients who do not have any ear pathology and undergo surgery under general anesthesia, on the MEP.

DETAILED DESCRIPTION:
Studies reported that inhalation agents are more likely to have impacts on the middle ear pressure compared to intravenous anesthetic agents. Despite numerous studies comparing the effects of inhalation agents on the middle ear pressure, this is the first clinical trial in which end tidal carbon dioxide and effects of sevoflurane and desflurane, along with other anesthetic analgesic agents used, on the middle ear pressure were compared. Our purpose in this study was to investigate the effect of sevoflurane and desflurane, inhalation agents used in patients who do not have any ear pathology and undergo non-ear surgery under general anesthesia, on the middle ear pressure.

ELIGIBILITY:
Inclusion Criteria:

* (ASA) II-III physical status
* elective inguinal hernia
* lower extremity surgery
* general anesthesia
* supine position

Exclusion Criteria:

* nasal septum,
* adenotonsillar hypertrophy,
* perforated tympanic membrane,
* middle ear pathology
* receive medications for middle ear pressure .

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2013-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Middle ear pressure | postoperative 30th minutes
  Tympanometric measurements were performed and recorded for each ear preoperatively, at intraoperative 5th, 10th and 15th minutes and postoperative 10th and 30th minutes. Normal middle ear pressure ranges between -200 and +200 decapascals (daPa).
  Treatment-Related Adverse Events, Ear and labyrinth disorder Assessed by CTCAE v4.0

IPD SHARING:
Plan to Share IPD: No